CLINICAL TRIAL: NCT02537548
Title: Surgery in Early Metastatic Seminoma (SEMS): Phase II Trial of Retroperitoneal Lymph Node Dissection as First-Line Treatment for Testicular Seminoma With Isolated Retroperitoneal Disease (1-3cm)
Brief Title: Retroperitoneal Lymph Node Dissection in Treating Patients With Testicular Seminoma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4T-14-1; NCI-2015-01177 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HS-15-00246; 4T-14-1 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2015-08-29; First posted 2015-09-01 (Estimated); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Lymphadenopathy; Stage I Testicular Seminoma; Stage II Testicular Seminoma
MeSH Terms: conditions — Lymphadenopathy; Seminoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (RPLND) (Experimental): Patients undergo RPLND.
  Interventions: Other: Laboratory Biomarker Analysis; Procedure: Retroperitoneal Lymph Node Dissection

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Retroperitoneal Lymph Node Dissection — Undergo RPLND
  Other Names: RPLND

SUMMARY:
This phase II trial studies how well retroperitoneal lymph node dissection (RPLND) works in treating patients with stage I-IIa testicular seminoma. The retroperitoneum is the space in the body behind the intestines that is typically the first place that seminoma spreads. RPLND is a surgery that removes lymph nodes in this area to treat testicular seminoma and may experience fewer long-term toxicities, such as a second cancer, cardiovascular disease, metabolic syndrome (pre-diabetes), or lung disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the recurrence free survival (RFS) at 2 years after RPLND when RPLND is used as a first line treatment for patients with testicular seminoma and low volume (=< 2cm) retroperitoneal disease.

SECONDARY OBJECTIVES:

I. Estimate the percent of patients, after treatment with RPLND, who can avoid external beam radiotherapy (XRT) or systemic chemotherapy (CTX) for seminoma.

II. Assess the complications associated with primary RPLND for seminoma.

OUTLINE:

Patients undergo RPLND.

After completion of study treatment, patients are followed up at 1 month, every 4 months for 1 year, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Pure seminoma after orchiectomy presenting with isolated retropreritoneal lymphadenopathy OR stage I pure seminoma with isolated retroperitoneal relapse. Relapse should be within 3 years
* Lymphadenopathy in the retroperitoneum: at least one lymph node 1-3 cm in greatest dimension, no lymph node > 3 cm in greatest dimension, no more than 2 lymph nodes 1-3 cm in greatest dimension

  * Axial imaging of lymphadenopathy within 6 weeks of the date of RPLND
  * Retroperitoneal lymphadenopathy must be within the RPLND template
* If there is borderline lymphadenopathy, defined as the largest retroperitoneal lymph node measuring 0.90 - 0.99 cm in the greatest dimension, an abdominal computed tomography (CT) scan should be repeated (recommend interval of 6 - 8 weeks); the same lymph node must demonstrate growth to >= 1.0 cm in the greatest dimension
* Biopsy is not required, though if biopsy of the retroperitoneal node(s) was obtained, pathology must be consistent with pure seminoma
* Chest imaging (x-ray, CT or magnetic resonance imaging [MRI]) negative for metastasis no more than 6 weeks prior to the date of RPLND
* Primary tumor excised by radical inguinal orchiectomy and pathology consistent with pure seminoma
* Serum alpha fetoprotein (AFP) not more than 1.5 times upper limit of normal, beta-human chorionic gonadotropin (HCG), lactate dehydrogenase (LDH) (per the local laboratory assay) within 14 days of RPLND
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Ability to understand and the willingness to sign a written informed consent
* Serum coagulation studies (INR/PTT) and platelet counts suitable for surgery per surgeon discretion.

Exclusion Criteria:

* Second primary malignancy
* History of receiving chemotherapy or radiotherapy
* Patients receiving any other investigational agent (s)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-08-28 (Actual); Primary Completion 2026-08-28 (Estimated); Study Completion 2027-08-28 (Estimated)

PRIMARY OUTCOMES:
RFS | From RPLND to the time of recurrence or death, whichever comes first., assessed at 2 years after RPLND
  Associated 95% confidence intervals will be constructed. Actuarial RFS will be calculated by the Kaplan Meier method. The recurrence location (pelvic, retroperitoneal, distant) will be calculated as a percentage of total recurrences to describe the clinical pattern of disease after relapse.

SECONDARY OUTCOMES:
Long-term RPLND complication rates | Up to 5 years
  The rate of short and long term complications will be calculated.
RFS | From RPLND to the time of recurrence or death, whichever comes first., assessed at 5 years after RPLND
  Associated 95% confidence intervals will be constructed. Actuarial RFS will be calculated by the Kaplan Meier method.
Short-term RPLND complication rates | Up to 12 months
  The rate of short and long term complications will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Siamak Daneshmand, Principal Investigator — University of Southern California
Locations (14):
- United States (14):
  - Loma Linda University Medical Center, Loma Linda, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Stanford University Hospitals & Clinics, Stanford, California
  - University of Colorado Hospital - Aurora, Aurora, Colorado
  - Emory University, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Stephenson Cancer Center, University of Oklahoma, Oklahoma City, Oklahoma
  - UTSouthwestern Medical Center, Dallas, Texas
  - Madigan Army Medical Center, Tacoma, Washington

REFERENCES:
- [Derived] Daneshmand S, Cary C, Masterson T, Einhorn L, Adra N, Boorjian SA, Kollmannsberger C, Schuckman A, So A, Black P, Bagrodia A, Skinner E, Alemozaffar M, Brand T, Eggener S, Pierorazio P, Stratton K, Nappi L, Nichols C, Luo C, Li M, Hu B. Surgery in Early Metastatic Seminoma: A Phase II Trial of Retroperitoneal Lymph Node Dissection for Testicular Seminoma With Limited Retroperitoneal Lymphadenopathy. J Clin Oncol. 2023 Jun 1;41(16):3009-3018. doi: 10.1200/JCO.22.00624. Epub 2023 Mar 13. PMID 36913642